CLINICAL TRIAL: NCT07373652
Title: Effects of Wrestling Training on Psychological Well-Being, Anxiety, and Resilience in Adolescent Boys
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gümüşhane Universıty (Other)
Responsible Party: Principal Investigator, Coşkun YILMAZ, ASSOC. PROF., Gümüşhane Universıty
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025/6
Record Dates: First submitted 2025-12-28; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Perceived Recovery
Keywords: psychological resilience; wellbeing; anxiety; mental health; adolescents; Wrestling
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study employed a randomized pretest-posttest control group design. Both groups underwent baseline assessments before the intervention and post-tests after six weeks. The Wrestling Group participated in a structured wrestling training program, while the Control Group maintained their usual daily routines without additional exercise. Participants visited the laboratory on three separate occasions. During the first visit, they were informed about the training protocol and completed familiarization procedures. The second visit (one week later) included baseline testing. The third visit occurred after the six-week intervention, during which all post-training assessments were conducted. All measurements were carried out under identical environmental conditions (temperature 22-24°C, relative humidity 45-55%) and supervised by the same research team to ensure consistency
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Wrestling Group (Experimental): The intervention consisted of a six-week wrestling training program conducted three times per week (Tuesday, Thursday, and Saturday) for 60 minutes per session
  Interventions: Other: Wrestling training; Other: Control
- CONTROL (No Intervention): Kontrol

INTERVENTIONS:
Other: Wrestling training — The intervention consisted of a six-week wrestling training program conducted three times per week (Tuesday, Thursday, and Saturday) for 60 minutes per session
  Arms: Experimental: Wrestling Group
Other: Control — Control
  Arms: Experimental: Wrestling Group

SUMMARY:
This study employed a randomized pretest-posttest control group design. Both groups underwent baseline assessments before the intervention and post-tests after six weeks. The Wrestling Group participated in a structured wrestling training program, while the Control Group maintained their usual daily routines without additional exercise. Participants visited the laboratory on three separate occasions. During the first visit, they were informed about the training protocol and completed the familiarization procedures. The second visit (one week later) included baseline testing. The third visit occurred after the six-week intervention, during which all post-training assessments were conducted. All measurements were carried out under identical environmental conditions (temperature 22-24°C, relative humidity 45%-55%) and supervised by the same research team to ensure consistency. The experimental flow is presented in Body composition measurement

DETAILED DESCRIPTION:
Materials and Methods Study design and Participants Thirty healthy male adolescents voluntarily participated in this randomized controlled study. Participants were randomly assigned to a Wrestling Group (WG; n = 15) or a Control Group (CG; n = 15) using an online randomization tool (www.randomizer.org). The required sample size was determined using the G*Power program (version 3.1.9.2; Düsseldorf, Germany). A power analysis revealed that at least 12 participants per group would be needed to identify statistically significant effects, with an effect size of 0.80 and actual power of 0.89, focusing on psychological resilience as the primary outcome measure. To account for possible dropouts, the sample size was increased by 25%, resulting in 15 participants per group (n = 30). Participants had to meet the inclusion criteria of being between 12-15 years of age, having no prior experience in wrestling or organized combat sports, and not having engaged in regular physical training for more than 60 minutes per week over the preceding six months. The exclusion criteria included any musculoskeletal injury, chronic illness, or psychological disorder that could interfere with participation. All participants and their parents were fully informed about the study's purpose and procedures, and written informed consent was obtained from the parents or legal guardians. The study protocol was approved by the Ethics Committee of Gümüşhane University (Approval No: 2025/6, June 25, 2025) and conducted in accordance with the principles of the Declaration of Helsinki.

Experimental design This study employed a randomized pretest-posttest control group design. Both groups underwent baseline assessments before the intervention and post-tests after six weeks. The Wrestling Group participated in a structured wrestling training program, while the Control Group maintained their usual daily routines without additional exercise. Participants visited the laboratory on three separate occasions. During the first visit, they were informed about the training protocol and completed the familiarization procedures. The second visit (one week later) included baseline testing. The third visit occurred after the six-week intervention, during which all post-training assessments were conducted. All measurements were carried out under identical environmental conditions (temperature 22-24°C, relative humidity 45%-55%) and supervised by the same research team to ensure consistency. The experimental flow is presented in Body composition measurement In the study, body composition (e.g., body fat percentage and muscle mass) was assessed using a Jawon Medical GAIA 359 Plus bioelectrical impedance analyzer (Jawon Medical Co., South Korea), with data managed through the BodyPass software (GAIA 359 Plus version). This device was used to confirm that all participants had comparable baseline body characteristics. Body weight was recorded using the same analyzer, while height (cm) was measured with a portable stadiometer (Seca 213, Seca GmbH & Co. KG, Hamburg, Germany).

Sport Anxiety Scale-2 (SAS-2) The Sport Anxiety Scale-2 (SAS-2) is a revised instrument originally developed to assess competitive anxiety in athletes. The updated version includes 15 items rated on a four-point Likert scale and provides a multidimensional view of anxiety symptoms related to sport performance. The Turkish adaptation and validation study by Akman et al. confirmed its reliability and construct validity for adolescent athletes. The scale measures three distinct aspects of competitive anxiety: worry, which refers to outcome-related and self-focused concerns; somatic anxiety, which reflects physiological tension and physical manifestations of stress; and concentration disruption, which describes difficulties in maintaining attentional focus during performance. Higher scores on each subdimension indicated more severe anxiety symptoms in that domain, and all items in this study were evaluated using a four-point response format ranging from "not at all" to "very much." The WHO-5 Well-Being Index The WHO-5 Well-Being Index is a brief and effective screening tool for assessing psychological well-being. The applicability study of the Turkish version of the WHO-5 was conducted by Eser et al. Participants were asked to indicate the extent to which each of the five statements has been true for them over the past 14 days. Items are scored on a scale from 0 (at no time) to 5 (all of the time), resulting in a total raw score ranging from 0 (absence of well-being) to 25 (maximal well-being). A standardized 100-point score can also be calculated by multiplying the raw score by four. The WHO-5 can also be used to monitor individual changes over time, with a score change of 10% or more (increase or decrease) considered clinically significant.

Brief Psychological Resilience Scale (BPRS) The Brief Psychological Resilience Scale (BPRS) was originally developed by Smith et al. to assess an individual's ability to recover from stress and maintain emotional balance, and it was later adapted for Turkish samples by Doğan [20]. The instrument consists of six items scored on a five-point Likert scale ranging from "strongly disagree" to "strongly agree," with three of the items (2, 4, and 6) reverse-coded. After adjustment of these items, the total scores may range from 6 to 30, where higher values represent greater psychological resilience. The BPRS offers a practical and time-efficient assessment method with demonstrated reliability and cultural applicability in the Turkish population [20]. In the current study, the internal consistency of the BPRS was found to be acceptable, with a Cronbach's alpha coefficient of 0.79.

Weekly training program The intervention consisted of a six-week wrestling training program conducted three times per week (Tuesday, Thursday, and Saturday), with each session lasting 60 minutes. Each session incorporated fundamental wrestling components, including basic stances and balance, mobility and entry techniques, contact and defensive fundamentals, strength and agility drills, technical integration, and combined practice sessions. Previous literature suggests that a training frequency of at least three sessions per week over six to twelve weeks is critical for achieving meaningful physical and neuromuscular adaptations. Therefore, a six-week program was deemed appropriate for this study.

The protocol was structured into three progressive phases under the supervision of three certified wrestling experts. Each session began with a 15-minute warm-up, including a five-minute low-intensity run followed by a 10-minute agility and coordination circuit (side steps, crossover steps, two-foot jumps, single-leg hops, squat jumps, high knees, lunges, cut kicks, and backward steps). This was followed by a five-minute dynamic stretching routine targeting the major muscle groups to enhance flexibility and reduce muscle stiffness.

The remaining 40 minutes constituted the main training phase, focusing on wrestling-specific drills integrating stances, mobility, contact and defensive techniques, as well as strength and agility exercises combined with technical applications to improve overall performance. All sessions were supervised to ensure correct execution and progression.

No injuries occurred during the intervention. All participants in the wrestling group completed the full program, attending all 18 scheduled sessions (100% adherence). Similarly, the control group completed all pre- and posttest assessments with no attrition.

Statistical analysis All statistical procedures were conducted using IBM SPSS Statistics (Version 21.0, Chicago, IL, USA). The level of significance was set at p < 0.05. The Shapiro-Wilk test was used to assess the normality of data distribution across variables. To examine the interaction between time (pre- and posttest) and group (wrestling vs. control), a two-way repeated-measures ANOVA was performed, followed-when appropriate-by Bonferroni-adjusted post hoc comparisons. Partial eta-squared (ηp²) values were also calculated to estimate effect size. In accordance with Richardson's guidelines, effect sizes were interpreted as small (ηp² ≈ 0.01), moderate (ηp² ≈ 0.06), or large (ηp² ≥ 0.14).

ELIGIBILITY:
Inclusion Criteria:

* were between 12-15 years of age
* had no previous experience in wrestling or organized combat sports
* had not engaged in regular physical training (> 60 minutes per week) during the previous six months.

Exclusion Criteria:

* Any musculoskeletal injury
* chronic illness
* psychological disorder that could interfere with participation.

Ages: 10 Years to 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2025-09-05 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Brief Psychological Resilience Scale - BPRS | 6 weeks
  The primary outcome is the change in total BPRS score to evaluate the effect of wrestling training on adolescents' ability to recover from stress and maintain emotional balance.

SECONDARY OUTCOMES:
Change in Psychological Well-Being (WHO-5 Well-Being Index) | 6 weeks
  To determine whether wrestling training improves overall psychological well-being as measured by the WHO-5 Index.
Change in Sport Anxiety (Sport Anxiety Scale-2 - SAS-2) | 6 weeks
  To assess changes in total sport anxiety and its subscales (worry, somatic anxiety, concentration disruption) following wrestling training.
Change in Body Composition Parameters (Body Fat %) | 6 weeks
  To confirm physical comparability and explore potential secondary physical effects of the intervention.
Change in Body Composition Parameters (Muscle Mass) | 6 Week
  To confirm physical comparability and explore potential secondary physical effects of the intervention.
Change in Body Composition Parameters (Weight) | 6 Week
  To confirm physical comparability and explore potential secondary physical effects of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: coşkun yılmaz, associate professor, Principal Investigator — Gümüşhane Universıty
Locations (1):
- Gumushane Univetsity, Gümüşhane, Kelkit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF